CLINICAL TRIAL: NCT03082911
Title: Effectiveness of a Brief Telephone Intervention to Improve Participation in a Colorectal Cancer Screening Program: a Randomized Controlled Trial
Brief Title: A Telephone Intervention to Improve Participation in a Screening Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Anna Selva, Medical doctor specialist in Preventive Medicine and Public Health, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Corporació Parc Taulí
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: screening; early detection; participation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone call (Experimental): A brief telephone intervention at the same time of sending the invitation letter plus the habitual invitation process used in the screening program (described in control group).
  Calls will be made by the administrative staff of the Screening Technical Office, which is experienced in telephone attention.
  Each phone call will last approximately 5 minutes.
  Interventions: Other: Phone call; Other: Invitation letter
- Standard procedure (Active Comparator): The habitual invitation strategy used in the screening program . Three letters are send by post: 1- An invitation letter plus an information leaflet and a list of pharmacies in which people can obtain the screening test. 2- A reminder letter for those who have not participated after 5 weeks of sending the first letter. 3- A second reminder letter for those who have collected the kit in the pharmacy but have not returned it with the sample.
  Interventions: Other: Invitation letter

INTERVENTIONS:
Other: Phone call — A brief telephone intervention at the same time of sending the invitation letter plus the habitual invitation process used in the screening program (described in control group). Each phone call will last approximately 5 minutes.
  Calls will be made by the administrative staff of the Screening Technical Office, which is experienced in telephone attention.
  Arms: Phone call
Other: Invitation letter — The habitual invitation strategy used in the screening program . Three letters are send by post: 1- An invitation letter plus an information leaflet and a list of pharmacies in which people can obtain the screening test. 2- A reminder letter for those who have not participated after 5 weeks of sending the first letter. 3- A second reminder letter for those who have collected the kit in the pharmacy but have not returned it with the sample

SUMMARY:
Objective: To assess the effectiveness of a brief telephone intervention added to an post invitation letter in the participation rate to a colorectal cancer screening program.

Methods: Randomized controlled trial. This study is framed inside the colorectal cancer screening program of Catalonia, concretely in the region of Vallès Occidental. This program is directed to men and women from 50 to 69 years. The screening test used is the fecal immunological test (FIT) that is offered every 2 years. If the screening test is positive, a colonoscopy with sedation is offered as a diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Women and men from 50 to 69 years living in the selected territories (Terrassa C, Terrassa A, Cerdanyola del Vallès 1) that will be invited for the first time in the Colorectal cancer screening program.

Exclusion Criteria:

* The same as those used in the population program:

  1. History of colorectal cancer;
  2. History of inflammatory bowel disease;
  3. history of colorectal adenomas;
  4. family history of polyposis syndromes or hereditary nonpolyposis colorectal cancer;
  5. family history of colorectal cancer if: two first grade relatives affected or only one fist grade relative affected diagnosed before the age of 60;
  6. terminal illness or severe disability which contraindicates the study of the colon. People is excluded temporally if:

     * 1) they have a colonoscopy performed in the last 5 years;
     * 2) present digestive signs or symptoms (rectal bleeding, change in bowel habits, abdominal pain, weight loss with fatigue and anorexia, abdominal mass);
     * 3) they express the will to be out of the Program.

Ages: 49 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Participation | 6 months
  Participation is defined as the number of people who do the screening test to the total of people invited to the Program.

SECONDARY OUTCOMES:
Knowledge of the program | 1 day at the time of intervention administration
  proportion of people from the intervention group who report knowing the existence of the program.
Comprehension of the information received | 1 day at the time of intervention administration
  proportion of people from the intervention group who report having understood in which the screening program consists of.
Help to decide about participation | 1 day at the time of intervention administration
  proportion of people from the intervention group who report that the information received in the phone call will be useful to decide about their participation in the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Selva A, Tora N, Pascual E, Espinas JA, Bare M. Effectiveness of a brief phone intervention to increase participation in a population-based colorectal cancer screening programme: a randomized controlled trial. Colorectal Dis. 2019 Oct;21(10):1120-1129. doi: 10.1111/codi.14707. Epub 2019 Jun 17. PMID 31099455